CLINICAL TRIAL: NCT07114705
Title: The Relationship Between the Number of Ceserean Sections and Scar Niche Development :Cross Sectional Study
Brief Title: The Relationship Between the Number of Ceserean Sections and Scar Niche Development
Status: Not yet recruiting | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Shimaa Nasser Ahmed, Resident doctor at obs gyna department sohag university, Sohag University
Other Study IDs: So-med-25-7-15MS
Record Dates: First submitted 2025-08-03; First posted 2025-08-11 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Scar Niche; Infertility, Post Menstrual Spotting
Keywords: Scar niche
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group 1: Women with 1 Previous Cesarean Section or more
  Interventions: Diagnostic Test: Transvaginal ultrasound

INTERVENTIONS:
Diagnostic Test: Transvaginal ultrasound — This is the only method

SUMMARY:
Aim of the work This study aims to investigate the relationship between the number of previous cesarean sections (CS) and the incidence of a cesarean scar niche.

DETAILED DESCRIPTION:
Cesarean section (CS) is a common surgical procedure globally, with increasing rates over the past few decades (WHO, 2021). This rise has led to concerns about its long-term complications, including the formation of Cesarean scar niches, also known as isthmoceles (the most common), Cesarean scar defect, Cesarean scar pouch, Cesarean scar diverticulum, Uterine niche and Myometrial defect at cesarean scar. These niches are characterized by discontinuation of the myometrium at the site of the previous CS, often presenting as a hypoechoic area within the lower uterine segment (Elkashef et al., 2023).

The prevalence of cesarean scar niches varies widely, ranging from 6.9% to 69%, depending on the diagnostic method used and the population studied (Elkashef et al., 2023; Alassi et al., 2022). In Egypt, the incidence of CS has increased significantly, contributing to a higher risk of niche formation. Recent studies have highlighted a significant relationship between the number of cesarean deliveries and the risk of developing a scar niche, with multiple CS being a major risk factor (Elkashef et al., 2023).

For instance, multiple cesarean sections may interfere with tissue perfusion and are associated with increased width and depth of the scar defects (Tilahun et al., 2023).

Cesarean scar niches are associated with various clinical symptoms, including abnormal uterine bleeding, chronic pelvic pain, dysmenorrhea, and subfertility, significantly impacting a woman's quality of life (Alassi et al., 2022). The formation of these niches can also lead to complications such as ectopic pregnancies and placenta accreta spectrum disorders (Jauniaux, et al., 2022). Understanding these risks and factors is crucial for developing preventive strategies and managing potential complications.

ELIGIBILITY:
Inclusion Criteria:

* History of at least one previous cesarean section in non pregnant women.

Exclusion Criteria:

* Women with known uterine anomalies (e.g., bicornuate uterus, uterine septum). Previous uterine surgery other than CS (e.g., myomectomy). History of uterine rupture in previous pregnancies.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Females
Study Population: The study population includes women of reproductive age who have undergone one or more cesarean section deliveries. Participants will be recruited from obstetrics and gynecology outpatient clinics. The study focuses on evaluating the presence and severity of scar niche in relation to the number of cesarean sections.
Sampling Method: Non-Probability Sample
Enrollment: 82 (Estimated)
Dates: Start 2025-08-02 (Estimated); Primary Completion 2026-08-02 (Estimated); Study Completion 2026-09-02 (Estimated)

PRIMARY OUTCOMES:
Name Presence of Cesarean Scar Niche | At time of ultrasound evaluation
  Detection of cesarean scar defect (niche) using transvaginal ultrasound.

IPD SHARING:
Plan to Share IPD: Undecided
I dont know